CLINICAL TRIAL: NCT02075177
Title: Expanded Access Study of Fenretinide (4-HPR, NSC 374551) Lym-X-Sorb (LXS) Oral Powder Plus Ketoconazole in Patients With Recurrent or Resistant Neuroblastoma (IND#68,254)
Brief Title: Expanded Access Study of Fenretinide Lym-X-Sorb Plus Ketoconazole in Neuroblastoma
Status: No longer available | Type: Expanded Access
Sponsor: South Plains Oncology Consortium (Network)
Responsible Party: Sponsor
Other Study IDs: SPOC-2014-001
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Neuroblastoma; Neuroblastoma
Keywords: neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Fenretinide; Ketoconazole

INTERVENTIONS:
Drug: Fenretinide Lym-X-Sorb Oral Powder — Fenretinide Lym-X-Sorb 1500 mg/m2/day, daily for 7 days every 3 weeks
  Other Names: 4-HPR; Fenretinide; 4-HPR/LXS; Fenretinide/LXS
Drug: Ketoconazole — Ketoconazole 6 mg/kg/day, daily for 7 days every 3 weeks.

SUMMARY:
Currently there is no known effective treatment for recurrent/resistant neuroblastoma.

Fenretinide is an anticancer agent that may work differently than standard chemotherapy medicines. It may cause the buildup of wax-like substances in neuroblastoma cancer cells, called "ceramides" or other chemicals, called 'reactive oxygen species'. In laboratory studies it was found that if too much ceramide or reactive oxygen species build up in neuroblastoma cells, they may die.

In addition, researchers are testing to see if a drug called ketoconazole, commonly used to treat fungus infections, can increase fenretinide levels in the body by interfering with the body's ability to break down fenretinide.

This study is being done: 1) to allow patients with recurrent/refractory neuroblastoma patients who would otherwise not be able to access fenretinide/LXS oral powder for treatment to do so; 2) to further describe the side effects of fenretinide and ketoconazole when given by mouth for seven days every three weeks; 3) to determine if a patient's tumor gets smaller after treatment with fenretinide oral powder plus ketoconazole or fenretinide oral powder alone.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of neuroblastoma either by histologic verification and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
* must have high risk neuroblastoma with one of the following: 1) recurrent/progressive disease at any time, 2) refractory disease, 3) persistent disease after at least a partial response to frontline therapy, or 4) Second or greater complete remission after definitive disease progression.
* must have at least one of the following sites of disease: 1) measurable tumor on MRI, CT scan, or X-Ray; 2)MIBG scan with positive uptake in at least one site; 3) bone marrow with tumor cells seen on routine morphology.
* must have an ECOG performance status of 0, 1, or 2
* must have a life expectancy of greater than or equal to 8 weeks
* must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* hemoglobin greater than or equal to 8.0 (may transfuse to achieve this level)
* ANC greater than or equal to 500 (must be at least 7 days after last dose of growth factor)
* platelet count greater than or equal to 50,000 (must be transfusion independent, defined as at least 1 week since last platelet transfusion)
* age-adjusted serum creatinine less than or equal to 1.5 times normal for age
* normal cardiac function documented by: ejection fraction (greater than or equal to 55%) documented by echocardiogram or radionuclide MUGA evaluation OR fractional shortening (greater than or equal to 27%) documented by echocardiogram AND EKG must demonstrate no abnormality severe enough to justify cardiac medications AND baseline QTc interval greater than or equal to 450 msecs
* total bilirubin less than or equal to 1.5 times normal for age
* ALT and AST less than or equal to 3 times normal for age (for this study, the upper limit of normal of ALT is defined as 45 U/L)
* normal prothrombin time (PT) for age
* baseline hepatitis titers without evidence of acute/active hepatitis. Patients will need to have a negative Hep B Surface Antigen (HBsAg), Hep B e Antigen (HBeAg), Anti-Hep B core Antibody IgM (Anti-HBc IgM), Anti-HAV IgM, and Anti-HCV IgM.
* Patients with CNS parenchymal or meningeal-based lesions are eligible. Patients with prior history of CNS irradiation are study eligible.
* Patients with a seizure disorder are eligible if seizures are controlled on anticonvulsants and if the specific anticonvulsant(s) is not contraindicated.
* Normal lung function as manifested by no dyspnea at rest and no oxygen requirement.
* Due to the potential teratogenic effects of retinoids, negative serum beta-HCG in females, and use of effective contraception in males and females of child-bearing potential, is required.
* skin toxicity no greater than grade 1 per CTCAE v4
* Serum triglycerides < 300mg/dL fasting or on a random plasma test.
* Serum calcium < 11.6mg/dL
* No hematuria and/or proteinuria greater than 1+ on urinalysis.
* Patients with known genetic metabolic conditions, or other ongoing serious medical issues, must be approved by the Study Chair prior to registration.

Exclusion Criteria:

* Pregnancy or breast feeding. Due to the potential teratogenic effects of retinoids, pregnant women are NOT eligible. Breast milk feeding by study patient is NOT allowed.
* Patients with history of organ and allogeneic stem cell transplantation.
* Patients with a known history of allergy to soy products.
* Patients with a known history of a severe allergy or sensitivity of wheat gluten.
* Patients requiring anti-arrhythmia cardiac medications are NOT eligible.
* Prior therapy with fenretinide, or fenretinide + ketoconazole, if DLT's were experienced.
* A known history of intolerance of ketoconazole.
* Patients on other essential medications for which an interaction with ketoconazole can be expected and for which dose reductions to other essential medications cannot be made in a manner adequate to ensure patient safety.
* Patients who, in the opinion of the investigator, may not be able to comply with safety monitoring requirements of the study.
* Active hepatitis.
* Baseline cardiac QTc interval >450 msecs.
* Eligible for enrollment on other national or regional treatment protocols employing fenretinide/LXS oral power that are reasonably accessible to the patient.
* Patient must NOT receive other anti-cancer agents while on Study.
* Ceftriaxone (Rocephin®) is NOT permitted for 24 hours prior to the start of the oral fenretinide course, during the course, and for 24 hours after the completion of seven day fenretinide course due to concerns of possible adverse effects on the hepatic clearance of fenretinide. Alternative antibiotics should be used. Other cephalosporins are permitted.
* Acetaminophen (Tylenol®) is NOT permitted for 24 hours prior the start of the oral fenretinide course, during the course, and for 48 hours following the completion of the seven day fenretinide course due to concerns of possible hepatic interactions. Ibuprofen (Motrin®) should be used for antipyretic control during this time period.
* Palliative radiation is allowed.
* Patients should NOT receive supplemental Vitamin A, C, or E except as contained in routine total parenteral nutrition vitamin supplements, or in a single daily standard dose oral multivitamin supplement, because of possible interference with antitumor 4-HPR-induced, reactive oxygen species and/or ceramide, and due to the unknown effects of these drugs on retinol levels
* Patients must NOT take any drugs suspected of causing pseudotumor cerebri, which include tetracycline, nalidixic acid, nitrofurantoin, phenytoin, sulfonamides (Dapsone permitted), lithium, amiodarone, or vitamin A (except as part of routine TPN supplements or as part of a single daily standard dose oral multivitamin supplement).
* Concomitant use of herbal supplements or other alternative therapy medications IS CONTRAINDICATED due to potential adverse metabolic interactions of such supplements with fenretinide.
* Patients should NOT concurrently take medications that may potentially act as modulators of intracellular ceramide levels or ceramide cytotoxicity, sphingolipid transport, or p-glycoprotein (MDR1) or MRP1 drug/lipid transporters, such as: cyclosporine A or analogue; verapamil; tamoxifen or analogue; chlorpromazine; RU486; indomethacin; or sulfinpyrazone. Patients should NOT concurrently take medications that are known P450 inhibitors. Contact Study Chair if there are questions regarding the suitability of any medication.
* As corticosteroids may impact sphingolipid metabolism, systemic corticosteroids should NOT be used for emesis control during the course of the study. Systemic corticosteroids for asthma control are permissible but should be minimized. Inhaled corticosteroids for asthma control are allowed. Steroids for routine metabolic deficiency states are allowed. Steroids for CNS lesions are allowed.
* Because gastric acidity is necessary for the maximal dissolution and absorption of ketoconazole, when actively taking ketoconazole, patients should avoid/minimize concurrent medications that decrease gastric acid output (such as ranitidine) or increase gastric pH (such as Tums).
* Concomitant medication that may prolong cardiac QT interval, especially those with known interaction with ketoconazole (See Appendices IV, V and VI). A LIST OF THESE MEDICATIONS SHOULD BE PROVIDED TO THE PATIENT AND FAMILY - PLEASE SEE APPENDICES IV, V and VI FOR A LIST OF MEDICATIONS THAT SHOULD NOT BE USED WITH CONCURRENT KETOCONAZOLE OR THAT SHOULD BE USED WITH CAUTION. Please SEE APPENDIX IV for a partial list of medications potentially prolonging QT interval. Patients may NOT receive therapy with the medications listed as PROHIBITED in Appendix IV and V. Medications in Appendix VI may be used with cautions as noted.

Regulatory:

* Patients and/or their parents or legal guardians must sign a written informed consent (or assent.)
* All institutional, FDA, and NCI requirements for human studies must be met.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - UT Southwestern Medical Center, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas